CLINICAL TRIAL: NCT06230211
Title: Effect of Maternal Voice and Music Therapy on Pain and Physiological Parameters During the Suction Procedure in Intubated Children: Randomized Controlled Study
Brief Title: Effect of Maternal Voice and Music Therapy on Pain and Physiological Parameters During in Intubated Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Fulya Kos, lecturer, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: BSEU-DEU
Record Dates: First submitted 2024-01-11; First posted 2024-01-30 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Music Therapy; Pain; Physiological Parameters; Mother's Voice
Keywords: Music Therapy; Mother's Voive
MeSH Terms: conditions — Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music therapy (Experimental): In the group where music therapy will be applied, the endotracheal aspiration and study to be performed will be explained to the child's family, and after obtaining consent, the music therapy applied to the child will be applied 5 minutes before, during and after the procedure. Meanwhile, the data will be recorded on the form by the observer. The song "The Happiest Child", developed by creating rhythms by Fulya Merve KOS, one of the researchers who has the RhythmotherapistTM certificate issued by the Ministry of National Education, will be used in music therapy. The sound will be adjusted to 45 db. The speaker will be placed at the end of the foot, approximately 30 cm from the child's ear, five minutes before the procedure and will be played to the child during the procedure.
  Interventions: Other: Music Therapy
- Mother's voice (Experimental): In the group where the mother's voice will be listened to, it will be explained to the child's parents that the mother's voice will be used for pain relief in the research. In the study, the researcher will take a voice from the mother of each child admitted to intensive care and record it on a voice recorder. Measurements will be made by placing the voice recorder 50 cm closer to the child to listen to the mother's voice. The volume of the mother's voice will be adjusted to an average of 45 decibels. The speaker will be placed at the end of the foot, approximately 30 cm from the child's ear, five minutes before the procedure and will be played to the child during the procedure.
  Interventions: Other: Maternal Voice

INTERVENTIONS:
Other: Music Therapy — Effect of Maternal Voice and Music Therapy on Pain and Physiological Parameters During the Suction Procedure in Intubated Children: Randomized Controlled Study
  Arms: music therapy
Other: Maternal Voice — Effect of Maternal Voice and Music Therapy on Pain and Physiological Parameters During the Suction Procedure in Intubated Children: Randomized Controlled Study
  Arms: Mother's voice

SUMMARY:
Children on mechanical ventilation are given painful stimuli an average of 10-14 times a day, and endotracheal aspiration is one of the procedures that causes the most pain in these children. Effective pain control not only improves the quality of life of children undergoing cardiothoracic surgery, but can also improve clinical outcome. If pain is not alleviated or eliminated with effective interventions during this period, it may cause neurological and behavioral disorders in the future. Excessive and long-term pain, especially as a result of applied interventions, causes behavioral stress and physiological imbalances. Any painful invasive procedure may interfere with the child's behavior, nutrition routine, interaction with the mother, and the child's adaptation to the environment, as well as may cause postoperative complications. In addition, experiencing pain can affect subsequent pain behaviors, causing the child to have a sensitivity to pain throughout his life. Effective pain management is divided into two categories: pharmacological and non-pharmacological. Non-pharmacological pain management strategies in children Pain management is defined as any strategy or technique applied to a child in pain with the aim of reducing the pain experience. Listening to recorded maternal voice and maternal heartbeat, music therapy, white noise are some of the non-pharmacological methods used in children. Studies emphasize that the use of music therapy is an effective method to reduce postoperative pain, ensure better oxygenation and improve physiological parameters in children who have undergone major surgery such as cardiothoracic surgery. It is also emphasized that music therapy reduces respiratory frequency, stabilizes breathing, stimulates the pituitary gland to secrete endorphins, and stabilizes heart rate and blood pressure by reducing catecholamine levels. It is stated that one of the non-pharmacological methods used in effective pain management in children is the mother's voice. Although the mechanism underlying the effect of the mother's voice is not fully explained, it is stated that the mother's voice will create a relaxing environment for children. Studies have shown that listening to the mother's voice before and after invasive interventions on babies and children in the intensive care unit reduces pain. In a study conducted by Erdoğan and his colleagues, they found that the pain levels, heart rates and oxygen saturations of children aged 1-3 who were listened to the mother's voice during painful procedures were lower. It is emphasized that listening to the mother's voice is one of the approaches that can be used as an effective method in pain management in critical care environments where mothers cannot be with their babies and children and cannot actively participate in their care.

It is known that non-pharmacological methods are effective in reducing pain in children, and they increase the effectiveness of drugs when used together with analgesics. Non-pharmacological methods are preferred because they are easy to apply and cheap, and they reduce the need for drug administration and thus the risk of side effects. Knowing the impact of pain and related stress on children, developing appropriate pain control strategies is both a medical and ethical responsibility. When the literature is examined, it is thought that there are a limited number of studies examining the effects of mother's voice and music therapy on pain and physiological parameters during the aspiration process in intubated children, and that not examining "mother's voice and music therapy", which directly affects pain and physiological parameters during the aspiration process in intubated children, is an important limitation. In this context, the aim of the study is to examine the effects of mother's voice and music therapy on pain and physiological parameters during the aspiration process in intubated children.

DETAILED DESCRIPTION:
Congenital heart disease (CHD) is defined as the most common congenital anomaly in the neonatal period, which refers to structural, functional or metabolic abnormalities of the heart or major blood vessels that occur during embryogenesis. It is stated that it is responsible for 28% of all major congenital anomalies. The incidence of congenital heart diseases, which is a chronic disease that requires lifelong follow-up, has been reported as 9.41/1,000 worldwide. In epidemiological studies conducted in our country, the incidence of congenital heart disease has been reported to be between 0.06-1.6%. According to the data of the Turkish Statistical Institute, it is stated that the number of babies born with congenital heart diseases every year in our country is 12,000-13,000. It is known that the most effective method used in the treatment of children with congenital heart disease is cardiothoracic surgery. The most common complication in children undergoing cardiothoracic surgery is pain. Studies have shown that 24-80% of children undergoing surgery are accompanied by moderate and severe pain. Cardiothoracic surgery is often completed with sternotomy or thoracotomy, and postoperative pain intensifies due to the long duration of the surgery and the damage to the chest muscles and nerves caused by the surgery. Studies have reported that pain increases by 10% in the first 24 hours after surgery, especially after the interventions. Children hospitalized in the intensive care unit after cardiothoracic surgery and especially those receiving mechanical ventilation are exposed to painful stimuli due to many procedures performed to monitor their vital signs and improve their physiological conditions. Children on mechanical ventilation are given painful stimuli an average of 10-14 times a day, and endotracheal aspiration is one of the procedures that causes the most pain in these children. After routine invasive procedures that cause pain, such as endotracheal aspiration, negative physiological, metabolic and behavioral responses may occur in children as stress, duration and severity of pain increase. Increases in heart rate, respiratory rate and blood pressure are observed due to catecholamines, glucagon and steroids released following painful stimuli, and these physiological changes observed in response to pain are thought to play a role in the initiation of ischemic changes by causing intraventricular bleeding and white matter damage around the ventricle. It is also reported that a baby who feels pain cannot adapt to the mechanical ventilator and mechanical ventilation becomes difficult. Pain that occurs after major surgery, especially invasive procedures, has a significant impact on the health status of children and should be intervened as early as possible. Effective pain control not only improves the quality of life of children undergoing cardiothoracic surgery, but can also improve clinical outcome. If pain is not alleviated or eliminated with effective interventions during this period, it may cause neurological and behavioral disorders in the future. Excessive and long-term pain, especially as a result of applied interventions, causes behavioral stress and physiological imbalances. Any painful invasive procedure may interfere with the child's behavior, nutrition routine, interaction with the mother, and the child's adaptation to the environment, as well as may cause postoperative complications. In addition, experiencing pain can affect subsequent pain behaviors, causing the child to have a sensitivity to pain throughout his life. Effective pain management is divided into two categories: pharmacological and non-pharmacological. Non-pharmacological pain management strategies in children Pain management is defined as any strategy or technique applied to a child in pain with the aim of reducing the pain experience. Listening to recorded maternal voice and maternal heartbeat, music therapy, white noise are some of the non-pharmacological methods used in children. It is stated that music therapy is one of the non-pharmacological methods commonly used in postoperative analgesia, which has effects that increase the release of endorphin hormone and reduce the need for analgesics by reducing catecholamine levels, stabilize heart rhythm and respiratory rate, maintain hemodynamic balance, affect the regional activity of the heart and reduce blood pressure. Studies emphasize that the use of music therapy is an effective method to reduce postoperative pain, ensure better oxygenation and improve physiological parameters in children who have undergone major surgery such as cardiothoracic surgery. It is also emphasized that music therapy reduces respiratory frequency, stabilizes breathing, stimulates the pituitary gland to secrete endorphins, and stabilizes heart rate and blood pressure by reducing catecholamine levels.

It is stated that one of the non-pharmacological methods used in effective pain management in children is the mother's voice. Although the mechanism underlying the effect of the mother's voice is not fully explained, it is stated that the mother's voice will create a relaxing environment for children. Studies have shown that listening to the mother's voice before and after invasive interventions on babies and children in the intensive care unit reduces pain. In a study conducted by Erdoğan and his colleagues, they found that the pain levels, heart rates and oxygen saturations of children aged 1-3 who were listened to the mother's voice during painful procedures were lower. It is emphasized that listening to the mother's voice is one of the approaches that can be used as an effective method in pain management in critical care environments where mothers cannot be with their babies and children and cannot actively participate in their care.

It is known that non-pharmacological methods are effective in reducing pain in children, and they increase the effectiveness of drugs when used together with analgesics. Non-pharmacological methods are preferred because they are easy to apply and cheap, and they reduce the need for drug administration and thus the risk of side effects. Knowing the impact of pain and related stress on children, developing appropriate pain control strategies is both a medical and ethical responsibility. When the literature is examined, it is thought that there are a limited number of studies examining the effects of mother's voice and music therapy on pain and physiological parameters during the aspiration process in intubated children, and that not examining "mother's voice and music therapy", which directly affects pain and physiological parameters during the aspiration process in intubated children, is an important limitation. In this context, the aim of the study is to examine the effects of mother's voice and music therapy on pain and physiological parameters during the aspiration process in intubated children.

ELIGIBILITY:
Sampling Inclusion Criteria:

* Children must be between the ages of 2 - 36 months
* Having Passed the Newborn Audiology Test
* Requiring endotracheal aspiration,
* The patient's hemodynamic parameters monitored on the monitor are stable,
* 2 hours have passed since the last painful attempt
* Children whose parents agreed to participate in the study were included in the study.

Exclusion Criteria from the Sample:

* Having an auditory disorder
* Lack of Parental Consent Form

Ages: 2 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-02-02 (Estimated); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Descriptive Information Form | one year
  The form prepared by the researchers in line with the literature consists of 19 questions including socio-demographic characteristics, information about the child's disease, and the parent's pain perception. This form will also record the child's physiological parameters (heart rate, arterial blood pressure, respiratory rate and oxygen saturation) during the painful procedure.
  (0-1 year old pulse: 80<pulse value<160, 1-3 years old pulse: 80<pulse value<130, The normal blood pressure limit for a 2-year-old child is 92/44 mmHg. oxygen saturation>95, Respiratory rate: 30 - 35 in newborn babies, 25-30 in 2-year-old children.)
FLACC (Face, Legs, Arms, Cry, Consolability) Pain Scale | one year
  The abbreviation FLACC consists of the initials of the words face, legs, activity, cry and consolability.The FLACC pain scale evaluates five behavioral domains (infant-child facial expression, leg mobility, activity, crying, and consolability) with scores ranging from 0 to 2 for each item. Min. 0 and max. 10 points can be collected. It is stated that as the score increases, the pain level increases, and as it decreases, there is less pain. In scoring, 0 points indicate no pain, 1-3 points indicate mild pain, 4-6 points indicate moderate pain, and 7-10 points indicate severe pain. The validity and reliability of the FLACC pain scale in our country was determined. This scale can be applied observationally by health professionals.

IPD SHARING:
Plan to Share IPD: No